CLINICAL TRIAL: NCT06943937
Title: An Exploratory Clinical Study of YTS109 Cell in Subjects With Refractory Disease Systemic Lupus Erythematosus
Brief Title: A Clinical Study of YTS109 Cell in R/R Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YTS109-005
Record Dates: First submitted 2025-04-16; First posted 2025-04-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Lupus Nephritis (LN); Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Lupus Nephritis; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YTS109 cell (Experimental): Subjects will receive YTS109 cell (1E6 STAR+T cell/kg or 2E6 STAR+T cell/kg) once in this study.
  Interventions: Drug: YTS109 cell injection

INTERVENTIONS:
Drug: YTS109 cell injection — Subjects will receive YTS109 Cell Injection(1E6 STAR+T cell/kg or 2E6 STAR+T cell/kg) once in this study.

SUMMARY:
This study evaluates the safety and efficacy of YTS109 cells in adults with refractory Lupus Nephritis (LN) and Systemic Lupus Erythematosus-Immune Thrombocytopenia (SLE-ITP). Approximately 36 patients aged 18-65 will receive a single infusion of YTS109 cells (1×10⁶-2×10⁶ cells/kg). The primary endpoint is observations of types, severity, and frequency of dose-limiting toxicities (DLTs) and adverse events (AEs). Secondary endpoints include the complete renal response (CRR) rate at week 12 in LN, and proportion of subjects achieving complete response (CR) or partial response (PR) at week 12 post-treatment in SLE-ITP. This single-arm, open-label trial will enroll patients across Beijing GoBroad Hospital in China.

DETAILED DESCRIPTION:
Background: Systemic lupus erythematosus (SLE) is characterized by multi-system and multi-organ involvement, recurrent flares and remissions, and the presence of numerous autoantibodies. LN and SLE-ITP are the most common and severe clinical manifestations of SLE. Recently, the therapeutic advancements have been made in the management of SLE. However, the patients with refractory SLE, particularly those complicated by LN and SLE-ITP, continue to face significant unmet clinical needs. CAR-T cell therapy has emerged as one of the innovative therapeutic modalities for autoimmune diseases, characterized by its controllable safety profile and durable therapeutic efficacy, warranting further clinical exploration and investigation in the future. YTS109 cell is a universal allogeneic STAR-T cell therapy targeting CD19, designed to efficiently eliminate B cells in patients with SLE and mitigate autoimmune responses. Design: This is a single-center, single-arm, prospective exploratory clinical trial designed to evaluate the safety profile, preliminary therapeutic efficacy, and pharmacokinetic/pharmacodynamic (PK/PD) characteristics of YTS109 cell therapy in patients with refractory SLE. Approximately 36 patients aged 18-65 will receive a single infusion of YTS109 cells (1×10⁶-2×10⁶ cells/kg). The primary endpoint is observations of types, severity, and frequency of dose-limiting toxicities (DLTs) and adverse events (AEs). This study was approved by the IRB of Beijing GoBroad Hospital (Approval Number: RP2025-013-002), All participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in this study:

1. Age ranges from 18 to 65 years old (including threshold), regardless of gender.
2. Meet the EULAR/ACR 2019 SLE Classification Criteri:

Cohort 1: Refractory Lupus Nephritis: Defined as failure to achieve remission after treatment with corticosteroids and ≥2 immunosuppressants (e.g., CTX, tacrolimus, MMF, cyclosporine) and/or biologics, with urine protein/creatinine ratio (UPCR ≥1.0 g/g) , and renal pathology requirement scriteria: ISN/RPS 2003 Class III/IV proliferative lupus nephritis (or combined with type V features) , with ≤50% glomerulosclerosis.

Cohort 2: Refractory Immune Thrombocytopenia: Requires treatment failure with: Failed treatment with at least 1 course of MP shock (1g for 3 days) or high- dose glucocorticosteroids (1mg/kg/d equivalent dose of glucocorticosteroids) in combination with 1 or more immunosuppressive agents. At least 2 consecutive routine blood tests for platelets less than 50×10^9/L and >30×10^9/L were performed prior to enrolment. other non-SLE causes of thrombocytopenia, such as infections, myelosuppression and hypersplenism, were excluded.

3. Essential Organ Function Criteria:

1. Bone marrow: Neutrophils ≥1×10^9/L (within 2 weeks, excluding granulocyte colony-stimulating factor use).

   Hemoglobin ≥60 g/L.
2. Liver: ALT/AST ≤3×ULN (disease-related elevations permitted). TBIL

   ≤1.5×ULN (disease-related elevations permitted).
3. Renal: CrCl≥30mL/min (Cockcroft-Gault formula, excluding acute declines).
4. Coagulation: INR/PT ≤1.5×ULN.
5. Cardiovascular: Hemodynamic stability. 4. Fertile females or males with partners of childbearing age must use medically approved contraception or abstain during and ≥12 months post- treatment. Negative serum HCG test (within 7 days pre-enrollment) for fertile females; non-lactating.

5. Voluntary participation with signed informed consent and compliance.

Exclusions Criteria:

Subjects who meet any of the following exclusion criteria will not be admitted to the study:

1. Severe drug allergies or hypersensitivity.
2. Uncontrolled/untreated infections (fungal, bacterial, viral, etc.).
3. CNS disorders (exceptions: epilepsy, psychosis, organic brain syndrome, cerebrovascular accident, encephalitis, CNS vasculitis).
4. Heart failure intolerance.
5. Congenital immunoglobulin deficiency.
6. Malignancy within 5 years (exceptions: localized cancers with negligible metastasis risk).
7. End-stage renal failure.
8. Subjects positive for: HBsAg / HBcAb with HBV DNA > detection limit; HCV Ab + HCV RNA; HIV Ab; Syphilis test.
9. Deep vein thrombosis/pulmonary embolism within 6 months pre- screening.
10. Severe mental illness/cognitive impairment.
11. Participation in other clinical trials within 3 months pre-screening.
12. Use of immunosuppressants (within 5 half-lives) or biologics (within 4 weeks) pre-screening.
13. Pregnancy/breastfeeding or planned conception.
14. Other researcher-determined ineligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days for DLT during the treatment assessment period, and observation AEs will be conducted up to 52 weeks post-treatment.
  1. Dose-limiting toxicity (DLT);
  2. Types, severity, and frequency of adverse events (AEs).

SECONDARY OUTCOMES:
Efficacy Evaluation in LN | The complete renal response (CRR) rate at week 12 in LN, and observation will be conducted up to 52 weeks post-treatment.
  The proportion of subjects who achieved complete renal response (CRR) at 12 weeks
Efficacy Evaluation in SLE-ITP | The proportion of subjects achieving complete response (CR) or partial response (PR) at week 12 post-treatment in SLE-ITP, and observation will be conducted up to 52 weeks post-treatment.
  The proportion of subjects achieving complete response (CR) or partial response (PR) at 12 weeks
Peak Plasma Concentration (Cmax) of YTS109 | These detections will be conducted up to 52 weeks post-treatment.
  To evaluate the metabolic characteristics of YTS109
Time to Peak (Tmax) of YTS109 | These detections will be conducted up to 52 weeks post-treatment.
  To evaluate the metabolic characteristics of YTS109
Area under the plasma concentration versus time curve (AUC) of YTS109 | These detections will be conducted up to 52 weeks post-treatment.
  To evaluate the metabolic characteristics of YTS109
PD parameters | These detections will be conducted up to 52 weeks post-treatment.
  Changes in B cells quantification and phenotypic in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No